CLINICAL TRIAL: NCT03808597
Title: Free Digital Health Education for Diseases of Public Health Importance (HIV, Tuberculosis and Taenia Solium Cysticercosis/Taeniosis) in Iringa, Tanzania
Brief Title: Digital Health Promotion in Iringa, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Sokoine University of Agriculture (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Christine Holst, Doctoral Research Fellow, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DigI
Record Dates: First submitted 2019-01-02; First posted 2019-01-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Tuberculosis; Cysticercosis; Tapeworm Pork
Keywords: digital health; digital health promotion; health promotion; disease prevention; HIV; Tuberculosis; Cysticercosis
MeSH Terms: conditions — HIV Infections; Tuberculosis; Cysticercosis; Taeniasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in this group will be exposed to digital health promotion. Please note that the participants are not randomly chosen, but stratified after the project villages. The participants in this group belong to the villages: Izazi and Migoli.
  Interventions: Other: Digital health promotion intervention
- Control group (No Intervention): The participants in this group will be not be exposed to digital health promotion, but the villages will receive the intervention after one year. Please note that the participants are not randomly chosen, but stratified after the project villages.
  The participants in this group belong to the villages: Kimande and Idodi.

INTERVENTIONS:
Other: Digital health promotion intervention — Digital health promition related to HIV, Tuberculosis and TSCT in a digital format.
  Arms: Intervention group

SUMMARY:
Increased health education has the potential to facilitate better use of health care services and to promote early treatment, thus it can strengthen the health care system, and ultimately reduce morbidity and mortality. In this study, we will develop and test the effect of digital health messages related to HIV, Tuberculosis (TB) and Taenia solium cysticercosis/taeniosis (TSCT) (the intervention diseases) in Migoli and Izazi (the intervention villages), in Iringa, Tanzania (TZ).

The intervention is planned as follows: A digital platform, providing the intervention villages with digital health messages related to the above-mentioned diseases, will be implemented in TZ in 2019. The platform will be accessible free of charge, through own devices and tablets based in the local Wi-Fi spots in the villages.

In the first part of this project, the doctoral research fellow will participate in developing the digital health messages, together with experts from the medical and teaching environments in Tanzania, Norway, Germany and USA.

The second part of the PhD-project consists of a cluster non-randomised controlled trial and semi-structured interviews in Tanzania. The digital health messages will be physically shown to the participants in the intervention group. The study is planned to investigate the knowledge related to the intervention diseases, before the intervention, immediately after exposure to the intervention, and at follow-up points throughout one year, after the intervention has been implemented. Semi-structured interviews with clients (users of the intervention) from each of the intervention villages are included, to explore the perception and reception of the intervention.

The baseline study and the immediate after survey will take place in Tanzania in Q1 2019, while the other follow-up studies and interviews (3, 6 and 12 months after baseline) will be undertaken throughout one year.

DETAILED DESCRIPTION:
Introduction This protocol is registered in Helseforsk, University of Oslo, and the project has been assessed by Norwegian Centre for Research Data (NSD), ref. number 59643. Ethical approval from the National Institute for Medical Research (NIMR), Tanzania, has been granted with the reference number NIMR/HQ/R.8a/Vol IX/2947.

The PhD-project consist of three work packages (WPs): WP1: A systematic review and meta-analysis, WP2: A cluster non-randomised controlled trial and WP3: Semi-structured interviews with clients in the intervention group. Only WP2 and WP3 are elaborated upon in this protocol.

The planned research project will be included as a health-research component in the Norwegian Government- and Norwegian Research Council- funded innovation project "Non-discriminating access for Digital Inclusion" (DigI). The project runs from January 2017 to September 2020. Altogether 11 partners from eight countries are collaborating on the project. Professor Josef Noll from the Dept. of Technology Systems (ITS), University of Oslo (UiO), is the project owner, and the doctoral research fellow's co- supervisor. Responsible for the health-research component and main supervisor of the doctoral research fellow, is Professor Dr. Andrea Winkler at the Institute of Health and Society, UiO. Head in TZ, is Dr. Bernard Ngowi (HIV/AIDS and TB specialist) from NIMR and Associate professor Helena Ngowi (TSCT specialist) from Sokoine University of Agriculture (SUA). Associate professor Maurice Isabwe from Dept. of Information and Communication Technology at University of Agder is head of developing the digital health messages. This study is thus multicentre with several institutions responsible for research.

In Tanzania, DigI will facilitate a digital health education platform, where digital health messages related to HIV / AIDS, Tuberculosis (TB) and Taenia solium cysticercosis/taeniosis (TSCT) will be transferred to the community; hereby called clients, defined by the World Health Organization (2017) as "members of the public that are potential or current users of health services, including promotion activities" .

The digital health messages will be accessible at a Wi-Fi spot in the local village close to the local health post. The digital health messages will also be shown face-to-face to each of the participants in the intervention group, by enumerators in the research team from SUA and the doctoral research fellow. The intervention will be available for all clients in the intervention villages, not only for the participants in the study described in this protocol.

The intervention will be maintained by NIMR Muhimbili Centre in Dar es Salaam during the first phase, but is going to be managed as a sustainable business model where a local sales man or woman is selling vouchers to access the World Wide Web. NIMR have close contact with the village authorities and health workers in the intervention villages, and will be alerted if the intervention for some reason is not functioning. The Wi-Fi network that provides the access to the digital health education platform, reaches within a radius of 50 meters, and is driven by a solar panel. This means that the intervention will be accessible even if the electricity locally shuts down.

Background and Rationale Today's education channels are changing, thus health education interventions must meet the target population at their own level of technology, and further do rely upon the characteristics of the technology available. A useful tool to deliver education and improve health seeking behaviour and health-related lifestyle decisions, is mobile technologies, because they make people more contactable. Health seeking behaviour may change after the target group has been exposed to adequate health messages that provide relevant information to the target population, , thus digital health information can contribute to prevention and management of diseases.

Digital health and digital health education Digital health is defined by World Health Organization (2016) as "The use of digital, mobile and wireless technologies to support the achievement of health objectives. Digital health describes the general use of information and communications technologies (ICT) for health and is inclusive of both mHealth (mobile health) and eHealth (electronic health)" . eHealth is defined by the WHO (2005) as "the cost-effective and secure use of information and communications technologies in support of health and health-related fields, including health-care services, health surveillance, health literature, and health education, knowledge and research" . mHealth is a component of eHealth, and commonly referred to as the use of mobile and wireless technologies for health. WHO (2011) defines it as: "medical and public health practice supported by mobile devices, such as mobile phones, patient monitoring devices, personal digital assistants (PDAs), and other wireless devices" .

Health behaviour change may reduce the burden of preventable disease and death around the world, "as health education covers the continuum from disease prevention and promotion of optimal health to the detection of illness to treatment, rehabilitation, and long-term care" .

The use of eHealth is now understood as central in order to provide more care and better care to more people, especially those most in need. A key part of the Sustainable Development Goal 3 relates to reaching people with the information they need in order to live healthier lives, and eHealth is regarded as a tool to reach the public with health messages and support, as well as encouraging clients to take active roles in their health and wellbeing (ibid).

The use of smart devices and mobile data services are rapidly changing, and it is likely that an increasingly part of the population in for example Sub-Saharan Africa will have access to both in the future.

ELIGIBILITY:
Inclusion Criteria:

* Living in the selected household (15-70 years), at least for the past six months, and at least planning to not move the next 12 months.
* Must be capable and willing to sign written informed consent and thumb-print for illiterate participants

Exclusion Criteria:

* Planning to be out of the village for more than 6 weeks in the next 12 months
* Those above 71 or under 15
* Not capable of signing consent letter (very sick)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Baseline Health knowledge score | One day
  Score calculated from the questionnaire with questions related to HIV, TB and TSCT. The score is calculated on the number of correct answers. The questionnaire contains 42 questions. If each question is correctly answered, the total score will be 225 (5 point for each question - weighted equally). Higher values represent a better outcome.
Change from Baseline Health knowledge score, immediately after exposure | One day
  Score calculated from the questionnaire with questions related to HIV, TB and TSCT. Comparison between baseline score and immediate post intervention score.
  The score is calculated on the number of correct answers. The questionnaire contains 42 questions. If each question is correctly answered, the total score will be 225 (5 point for each question - weighted equally). Higher values represent a better outcome.
Change from Baseline Health knowledge score at 3 months | Up to 3 months
  Score calculated from the questionnaire with questions related to HIV, TB and TSCT. Comparison between baseline score and post intervention (3 months) score.
  The score is calculated on the number of correct answers. The questionnaire contains 42 questions. If each question is correctly answered, the total score will be 225 (5 point for each question - weighted equally). Higher values represent a better outcome.
Change from Baseline Health knowledge score at 6 months | Up to 6 months
  Score calculated from the questionnaire with questions related to HIV, TB and TSCT. Comparison between baseline score and post intervention (6 months) score.
  The score is calculated on the number of correct answers. The questionnaire contains 42 questions. If each question is correctly answered, the total score will be 225 (5 point for each question - weighted equally). Higher values represent a better outcome.
Change from Baseline Health knowledge score at 12 months | Up to 12 months
  Score calculated from the questionnaire with questions related to HIV, TB and TSCT. Comparison between baseline score and post intervention (12 months) score.
  The score is calculated on the number of correct answers. The questionnaire contains 42 questions. If each question is correctly answered, the total score will be 225 (5 point for each question - weighted equally). Higher values represent a better outcome.

SECONDARY OUTCOMES:
Participants own perspectives on the intervention (qualitative) | One hour
  In order to get complimentary qualitative data, 8-10 semi-structured interviews with clients from the intervention villages will be conducted. The main aim is to get people to reveal their own perspectives related to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea S Winkler, M, PhdD, Study Chair — University of Oslo
Locations (6):
- Tanzania (6):
  - National Institute for Medical Research / Muhimbili University, Dar es Salaam, Dar
  - Idodi, Iringa
  - Izazi, Iringa
  - Kimande, Iringa
  - Migoli, Iringa
  - Sokoine University of Agriculture, Morogoro

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: 2020

REFERENCES:
- [Derived] Holst C, Stelzle D, Diep LM, Sukums F, Ngowi B, Noll J, Winkler AS. Improving Health Knowledge Through Provision of Free Digital Health Education to Rural Communities in Iringa, Tanzania: Nonrandomized Intervention Study. J Med Internet Res. 2022 Jul 28;24(7):e37666. doi: 10.2196/37666. PMID 35900820
- [Derived] Holst C, Sukums F, Ngowi B, Diep LM, Kebede TA, Noll J, Winkler AS. Digital Health Intervention to Increase Health Knowledge Related to Diseases of High Public Health Concern in Iringa, Tanzania: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Apr 22;10(4):e25128. doi: 10.2196/25128. PMID 33885369
- See also: Research project site University of Oslo — https://www.med.uio.no/helsam/english/research/projects/free-digital-health-information-tanzania/index.html
- See also: Overarching project site — https://its-wiki.no/wiki/DigI:Home

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03808597/Prot_SAP_000.pdf